CLINICAL TRIAL: NCT06074913
Title: Early Warning of Diabetic Peripheral Neuropathy by Using Infrared Thermography and the Effectiveness of Electroacupuncture in Its Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Chinese Medical University (Other Government)
Responsible Party: Principal Investigator, Jianqiao Fang, professor, Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GZY-ZJ-KJ-23021-02
Record Dates: First submitted 2023-09-21; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetic Peripheral Neuropathy; Diabetes; Electroacupuncture
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy group (Other): After the healthy volunteers met the requirements through screening (i.e., demographic data recording,medical history taking, physical examination report review and recording on the day of enrollment), IRT was performed on the extremities, with 1 image automatically taken every 10 s for 1 min, and 6 images for each site.
  Interventions: Other: infrared thermography (IRT)
- Diabetic group (Other): After screening to meet the inclusion criteria for this study, IRT was performed on the extremities, with 1 image automatically taken every 10s for 1 min, and 6 images for each site.
  Interventions: Other: infrared thermography (IRT)
- Diabetic peripheral neuropathy group (Other): After screening to meet the inclusion criteria for this study, IRT was performed on the extremities, with 1 image automatically taken every 10s for 1 min, and 6 images for each site.
  Interventions: Other: infrared thermography (IRT)
- EA group (Experimental): Subjects in this group received electroacupuncture along with the basic treatment at a frequency of 2 treatments per week for 6 weeks for a total of 12 interventions.
  Interventions: Procedure: Basal therapy+EA
- Waiting list group (Other): The subjects in this group will receive only basal treatment with no additional therapies during the study period.
  Interventions: Other: Basal therapy

INTERVENTIONS:
Other: infrared thermography (IRT) — Temperatures and infrared thermograms were recorded in the region of the extremities of three groups of subjects by using an infrared thermographic camera.
  Arms: Diabetic group; Diabetic peripheral neuropathy group; Healthy group
Procedure: Basal therapy+EA — After specialist treatment, blood glucose is managed through hypoglycemic medications or insulin. Patients with both hypertension and hyperlipidemia are prescribed antihypertensive and lipid-lowering drugs. Additional medications are determined based on the patient's current medication regimen. 2. Acupoints: Qihai (RN6), Guanyuan (RN4), Xuehai (SP10), Yanglingquan (GB34), Zusanli (T36), Yinlingquan (SP9), Sanyinjiao (SP6), Xuanzhong (GB39), Jiexi (ST41), Zulinqi (GB41), Taichong (SP41). The electrode will be connected Yanglingquan (GB34) and Sanyinjiao (SP6), electrode wire will be connected to the electro-acupuncture apparatus using continuous wave with a frequency of 2Hz at an intensity suitable for the comfort of the subject.
  Arms: EA group
Other: Basal therapy — After specialist treatment, blood glucose is managed through hypoglycemic medications or insulin. Patients with both hypertension and hyperlipidemia are prescribed antihypertensive and lipid-lowering drugs. Additional medications are determined based on the patient's current medication regimen.
  Arms: Waiting list group

SUMMARY:
Part Ⅰ:Infrared thermograms of four parts of the soles of the feet, dorsum of the feet, palms of the hands, and dorsum of the hands of healthy volunteers, diabetic patients, and patients with diabetic peripheral neuropathy were collected by using infrared thermography, and the patterns of change in the average temperatures of the parts of the participants in the three groups were analysed and compared by using the accompanying software.

Part Ⅱ: Diabetic Peripheral Neuropathy (DPN) mainly presents with symmetrical pain,numbness, and ankylosing sensation, but reversal after diagnosis is particularly difficult. Electroacupuncture can significantly improve the function of peripheral nerves, regulate local blood flow, and reduce the inflammatory response to promote nerve regeneration, but no study has shown that electroacupuncture can effectively prevent the occurrence of DPN. Therefore, it is of great research significance to determine whether electroacupuncture has the possibility in preventing the occurrence of DPN.

DETAILED DESCRIPTION:
Part Ⅰ: We analyse and compare the change rules of average temperature in each area of the three groups of patients, explore the correlation between the temperature in each area of mild DPN patients and the duration of the disease, age, BMI, etc., and explore the optimal prediction threshold for the occurrence of DPN, as well as its sensitivity and specificity.

Part Ⅱ: A total of 50 diabetic subjects meeting the inclusion criteria will be enrolled in the study and randomised into the EA group and the waiting list group using envelope randomisation. The indexes of main outcome evaluation are: change in regional temperature. The indexes of secondary outcome evaluation are: 1) sensory nerve amplitude and conduction velocity (SNCV) of the tibial and peroneal nerves of the lower extremities, and motor nerve amplitude and conduction velocity (MNCV). 2) change in TCSS score, and 3) laboratory tests (glycated haemoglobin, fasting blood glucose, and postprandial 2h blood glucose). This study will evaluate the effectiveness of EA in preventing DPN.

ELIGIBILITY:
Inclusion Criteria:

* Part Ⅰ：

Inclusion criteria for healthy subjects:

1. Routine physical examination by the investigator to confirm the absence of heart and lung diseases, and the absence of serious underlying diseases such as digestive, urinary, haematological, endocrine, and neurological systems;
2. 18 years old ≤ age ≤ 85 years old, gender is not limited;
3. Have normal communication ability;
4. Those who have a sense of autonomy and independence, voluntarily submit to the study protocol and sign the informed consent form.

Inclusion criteria for diabetic patients

1. 18 ≤ age ≤ 85 years old, with any disease duration and any gender;
2. Lower limb nerve electromyography shows no slowing of conduction velocity;
3. Normal communication ability;
4. No serious heart, brain, liver, kidney and other internal diseases, no serious mental illness and cognitive impairment;
5. Those who have a sense of autonomy and independence, voluntarily submit to the study protocol, and sign the informed consent form.

Inclusion criteria for mild DPN patients

1. 18 years ≤ age ≤ 85 years with any disease duration and any gender;
2. Clear history of diabetes mellitus;
3. Lower limb nerve EMG showing reduced conduction velocity, and/or persistent pain and/or sensory abnormalities in the extremities (at least in both lower limbs), diminished ankle reflexes bilaterally or unilaterally, and diminished vibration sensation;
4. TCSS score of 6-8;
5. Have normal communication skills;
6. No serious heart, brain, liver, kidney and other medical disorders, no serious mental illness and cognitive impairment;
7. Those who have a sense of autonomy and independence, voluntarily submit to the study protocol, and sign the informed consent form.

   * Part Ⅱ：

Inclusion Criteria:

1. 18 years ≤ age ≤ 85 years with any disease duration and any gender;
2. Those with changes in thermal characteristics for early warning of DPN patients according to Part Ⅰ; (3) Those whose lower limb neuromuscular electromyography shows no slowing of conduction velocity; (4) Those with normal communication skills; (5) No serious heart, brain, liver, kidney and other internal diseases, no serious mental illness and cognitive impairment; (6) Have a sense of autonomy and independence, voluntarily submit to the study protocol, and sign the informed consent form.

Exclusion Criteria:

* Part Ⅰ： Exclusion criteria for healthy subjects

  1. Those with severe mental illness, depression, alcohol dependence, or a history of substance abuse;
  2. Volunteers who are in preparation for pregnancy, pregnant or breastfeeding;
  3. Volunteers who are participating in other interventional clinical trials;
  4. Those who have scars, hyperpigmentation, redness, swelling and heat pain on the skin at the testing site, thus affecting the accuracy of the test.

Exclusion criteria for diabetic patients

1. Persons with severe mental illness, depression, alcohol dependence, or a history of substance abuse;
2. Volunteers who are in preparation for pregnancy, pregnant or breastfeeding;
3. Those with acute complications such as combined diabetic ketoacidosis, peripheral neuropathy, lactic acidosis, and severe infections;
4. Volunteers who are participating in other interventional clinical trials;
5. Those who have scars, hyperpigmentation, redness, swelling and heat pain on the skin at the testing site, thus affecting the accuracy of the test.

Exclusion criteria for mild DPN patients

1. TCSS score > 8;
2. Those with peripheral neuropathy, ulcers and gangrene of the extremities due to various other causes (e.g., hypothyroidism, alcohol, drugs, heredity, etc.) or those with a history of skin ulceration or lesions that do not heal easily;
3. Women who are in preparation for pregnancy, during pregnancy, or breastfeeding;
4. Those with acute complications such as combined lactic acidosis and severe infections;
5. Those who suffer from serious liver or kidney damage or serious cardiovascular diseases and cannot take care of themselves;
6. Those who have scars or pigmentation on the skin at the testing site, which affects the accuracy of the test;

   * Part Ⅱ：

Exclusion Criteria:

(1) Those with severe mental illness, depression, alcohol dependence, or a history of substance abuse; (2) Volunteers who are in preparation for pregnancy, pregnant or breastfeeding; (3) Those with acute complications such as combined diabetic ketoacidosis, diagnosed DPN, lactic acidosis, and severe infections; (4) Those with no change in thermal characteristics for early warning of DPN patients according to the results of the Part Ⅰ; (5) Those with liver or kidney damage or cardiovascular diseases (angina pectoris, myocardial infarction, multiple cerebral infarction, cerebral haemorrhage, etc.) resulting in severe sequelae; (6) Volunteers who are participating in other interventional clinical trials; (7) Those who have scars, hyperpigmentation, redness, swelling and heat pain on the skin at the testing site, thus affecting the accuracy of the test.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Temperature of the soles of the feet | Baseline, 6 weeks
  Participants in part 1 and part 2 were tested, but participants in part 1 were tested only once at enrolment and patients in part 2 were tested once before and once after treatment.
Temperature of the instep | Baseline, 6 weeks
  Participants in part 1 and part 2 were tested, but participants in part 1 were tested only once at enrolment and patients in part 2 were tested once before and once after treatment.
Temperature of the palm | Baseline, 6 weeks
  Participants in part 1 and part 2 were tested, but participants in part 1 were tested only once at enrolment and patients in part 2 were tested once before and once after treatment.
Temperature of the back of the hand | Baseline, 6 weeks
  Participants in part 1 and part 2 were tested, but participants in part 1 were tested only once at enrolment and patients in part 2 were tested once before and once after treatment.

SECONDARY OUTCOMES:
Electromyogram examination-Sensory conduction velocity of superficial peroneal nerve | Baseline, 6 weeks
  Participants in part 1 （except Health Volunteers）and part 2 were tested, but participants in part 1 were tested only once at enrolment and patients in part 2 were tested once before and once after treatment.
Electromyogram examination-Sensory conduction velocity of sural nerve | Baseline, 6 weeks
  Participants in part 1 （except Health Volunteers）and part 2 were tested, but participants in part 1 were tested only once at enrolment and patients in part 2 were tested once before and once after treatment.
Electromyogram examination-Motor conduction velocity of Peroneal nerve | Baseline, 6 weeks
  Participants in part 1 （except Health Volunteers）and part 2 were tested, but participants in part 1 were tested only once at enrolment and patients in part 2 were tested once before and once after treatment.
Electromyogram examination-Motor conduction velocity of tibial nerve | Baseline, 6 weeks
  Participants in part 1 （except Health Volunteers）and part 2 were tested, but participants in part 1 were tested only once at enrolment and patients in part 2 were tested once before and once after treatment.
Toronto clinical scoring system | Baseline, 6 weeks
  Participants in part 1 （except Health Volunteers）and part 2 were tested, but participants in part 1 were tested only once at enrolment and patients in part 2 were tested once before and once after treatment.
  The scale is an assessment of foot sensation and has a total score of 19, divided into three sections: symptom score of 6, reflex score of 8 and sensory score of 5. Symptom score: 0 = absent, 1 = present; reflex score: 0 = normal, 1 = diminished, 2 = absent; sensory score: 0 = normal, 1 = abnormal.
Glycated haemoglobin (HbA1c) | Baseline, 6 weeks
  Participants in part 1 （except Health Volunteers）and part 2 were tested, but participants in part 1 were tested only once at enrolment and patients in part 2 were tested once before and once after treatment.
Fasting blood glucose (FPG) | Baseline, 6 weeks
  Participants in part 1 （except Health Volunteers）and part 2 were tested, but participants in part 1 were tested only once at enrolment and patients in part 2 were tested once before and once after treatment.
2-hour postprandial blood glucose (2hPG) | Baseline, 6 weeks
  Participants in part 1 （except Health Volunteers）and part 2 were tested, but participants in part 1 were tested only once at enrolment and patients in part 2 were tested once before and once after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiao Fang, Principal Investigator — The Third Clinical Medical College of Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hanzhou, Zhejiang, China

REFERENCES:
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] Li Y, Teng D, Shi X, Qin G, Qin Y, Quan H, Shi B, Sun H, Ba J, Chen B, Du J, He L, Lai X, Li Y, Chi H, Liao E, Liu C, Liu L, Tang X, Tong N, Wang G, Zhang JA, Wang Y, Xue Y, Yan L, Yang J, Yang L, Yao Y, Ye Z, Zhang Q, Zhang L, Zhu J, Zhu M, Ning G, Mu Y, Zhao J, Teng W, Shan Z. Prevalence of diabetes recorded in mainland China using 2018 diagnostic criteria from the American Diabetes Association: national cross sectional study. BMJ. 2020 Apr 28;369:m997. doi: 10.1136/bmj.m997. PMID 32345662
- [Background] Iqbal Z, Azmi S, Yadav R, Ferdousi M, Kumar M, Cuthbertson DJ, Lim J, Malik RA, Alam U. Diabetic Peripheral Neuropathy: Epidemiology, Diagnosis, and Pharmacotherapy. Clin Ther. 2018 Jun;40(6):828-849. doi: 10.1016/j.clinthera.2018.04.001. Epub 2018 Apr 30. PMID 29709457
- [Background] Bagavathiappan S, Saravanan T, Philip J, Jayakumar T, Raj B, Karunanithi R, Panicker TM, Korath MP, Jagadeesan K. Infrared thermal imaging for detection of peripheral vascular disorders. J Med Phys. 2009 Jan;34(1):43-7. doi: 10.4103/0971-6203.48720. PMID 20126565
- [Background] Lahiri BB, Bagavathiappan S, Jayakumar T, Philip J. Medical applications of infrared thermography: A review. Infrared Phys Technol. 2012 Jul;55(4):221-235. doi: 10.1016/j.infrared.2012.03.007. Epub 2012 Apr 13. PMID 32288544
- [Background] Zhou Q, Qian Z, Wu J, Liu J, Ren L, Ren L. Early diagnosis of diabetic peripheral neuropathy based on infrared thermal imaging technology. Diabetes Metab Res Rev. 2021 Oct;37(7):e3429. doi: 10.1002/dmrr.3429. Epub 2021 Feb 4. PMID 33307598
- [Background] Selvarajah D, Kar D, Khunti K, Davies MJ, Scott AR, Walker J, Tesfaye S. Diabetic peripheral neuropathy: advances in diagnosis and strategies for screening and early intervention. Lancet Diabetes Endocrinol. 2019 Dec;7(12):938-948. doi: 10.1016/S2213-8587(19)30081-6. Epub 2019 Oct 14. PMID 31624024
- [Background] Yu B, Li M, Huang H, Ma S, Huang K, Zhong Z, Yu S, Zhang L. Acupuncture treatment of diabetic peripheral neuropathy: An overview of systematic reviews. J Clin Pharm Ther. 2021 Jun;46(3):585-598. doi: 10.1111/jcpt.13351. Epub 2021 Jan 28. PMID 33511675
- [Background] Zhang R, Lao L, Ren K, Berman BM. Mechanisms of acupuncture-electroacupuncture on persistent pain. Anesthesiology. 2014 Feb;120(2):482-503. doi: 10.1097/ALN.0000000000000101. PMID 24322588